CLINICAL TRIAL: NCT02083744
Title: A Self-Care Intervention for Hispanic Patients With Heart Failure
Brief Title: Project Fluido: Fluid Watchers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10-05030; 69344 (Other: Robert Wood Johnson Foundation)
Record Dates: First submitted 2014-02-25; First posted 2014-03-11 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Self-care; Spanish
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Usual care group - patients will receive scales to take home and heart failure literature for self-monitoring of heart failure. Patients will complete final questionnaires
  Interventions: Behavioral: Usual Care
- Psychoeducational Counseling (Experimental): 1-on-1 psychoeducation session conducted by a bilingual research nurse at the clinic site or in the patient's home. Patients will receive a scale to measure weight, a diary to record weight and symptoms of heart failure, and telephone follow-up from the research nurse to reinforce the content of the education program every other week.
  Focus-groups - Perception of the intervention will be assessed with two focus groups.
  Interventions: Behavioral: PsychoEducational Support

INTERVENTIONS:
Behavioral: PsychoEducational Support
  Arms: Psychoeducational Counseling
Behavioral: Usual Care — Standard Heart Failure Care
  Arms: Control Group

SUMMARY:
The long-term goal of this research is to determine whether a psychoeducational intervention will support self-care behaviors in Hispanic patients with heart failure. The specific goal of this study is to determine whether a culturally-appropriate psychoeducational intervention in Hispanic patients with heart failure, compared to a control group, will improve heart failure knowledge and self-care behaviors.

We hypothesize that patients who receive the intervention will have improved heart failure self-care behaviors and depression scores as measured by the Self-Care Heart Failure Index and Patient Health Questionnaire.

DETAILED DESCRIPTION:
A randomized clinical trial research design is planned. Investigators will obtain baseline and final measures on the intervention and control groups. A sample of 60 adult Hispanic heart failure patients will be recruited. Each patient will either participate in the psychoeducational intervention or usual care. A repeated measures (longitudinal) analysis will be used to examine these aims by employing a linear mixed models approach. The basic analysis has one between subjects (fixed) factor, group, with 2 levels (education and control) and one repeated factor, time, with 2 levels (baseline and 12 months). This analysis allows for testing the main effect of group, main effect of time, and the group by time interaction. The potential benefit of improving heart failure knowledge and self-care in Hispanic heart failure patients is that these patients may better understand how to care for themselves. This study will provide data to examine the longer-term outcomes of emergency department visits and hospitalization events in Hispanic patients.

ELIGIBILITY:
Inclusion Criteria:

* have been hospitalized for heart failure within the previous 24 months
* identify themselves as Hispanic in origin
* speak and write in Spanish or English

Exclusion Criteria:

* live in a nursing home or institution,
* age less than 18
* cognitive deficits
* serious life-limiting co-morbidity such as active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12-22 (Actual); Study Completion 2014-12-22 (Actual)

PRIMARY OUTCOMES:
the Self-Care Heart Failure Index | 3 months
  Self-Care maintenance, management and confidence will be measured.

SECONDARY OUTCOMES:
Depression as measured by the Patient Health Questionnaire. | 3 months
  The Patient Health Questionnaire will screen for depression symptoms.

OTHER OUTCOMES:
Anxiety as measured by the Symptom Inventory Questionnaire | 3 months
  A questionnaire will be used to measure symptoms of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jill N Howie-Esquivel, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States